CLINICAL TRIAL: NCT03885934
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of Catch-up Vaccination Regimens of V114 in Healthy Infants, Children, and Adolescents (PNEU-PLAN)
Brief Title: Safety and Immunogenicity of Catch-up Vaccination Regimens of V114 (V114-024)
Acronym: PNEU-PLAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-024; 2018-003706-88 (EudraCT Number)
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- V114, Schedule A: Participants 7-11 months (Experimental): Each participant received a 0.5 mL intramuscular (IM) injection for 7 to 11 months of age (Pneumococcal conjugate vaccine [PCV]-naïve)(3 doses). Dose 1: at randomization, Dose 2: 4 to 8 weeks after Dose 1, and Dose 3: 8 to 12 weeks after Dose 2 and ≥12 months of age.
  Interventions: Biological: V114
- Prevnar 13®, Schedule A: Participants 7-11 months (Active Comparator): Each participant received a 0.5 mL IM injection for 7 to 11 months of age (PCV-naïve)(3 doses). Dose 1: at randomization, Dose 2: 4 to 8 weeks after Dose 1, and Dose 3: 8 to 12 weeks after Dose 2 and ≥12 months of age.
  Interventions: Biological: Prevnar 13®
- V114, Schedule B: Participants 12-23 months (Experimental): Each participant received a 0.5 mL IM injection for 12 to 23 months of age (PCV-naïve)(2 doses). Dose 1: at randomization, and Dose 2: 8 to 12 weeks after Dose 1.
  Interventions: Biological: V114
- Prevnar 13®, Schedule B: Participants 12-23 months (Active Comparator): Each participant received a 0.5 mL IM injection for 12 to 23 months of age (PCV-naïve)(2 doses). Dose 1: at randomization, and Dose 2: 8 to 12 weeks after Dose 1.
  Interventions: Biological: Prevnar 13®
- V114, Schedule C: Participants 2-17 years (Experimental): Each participant received a 0.5 mL IM injection for 2 to 17 years of age (PCV-naïve or PCV-experienced) (1 dose). Single dose administered at randomization and at least 8 weeks after previous PCV for participants who were PCV-experienced.
  Interventions: Biological: V114
- Prevnar 13®, Schedule C: Participants 2-17 years (Active Comparator): Each participant received a 0.5 mL IM injection for 2 to 17 years of age (PCV-naïve or PCV-experienced)(1 dose). Single dose administered at randomization and at least 8 weeks after previous PCV for participants who were PCV-experienced.
  Interventions: Biological: Prevnar 13®

INTERVENTIONS:
Biological: V114 — V114 15-valent PCV containing 13 serotypes present in Prevnar 13® (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) and 2 unique serotypes (22F and 33F) in each 0.5 mL IM administration
  Other Names: Pneumococcal 15-valent Conjugate Vaccine, VAXNEUVANCE™
  Arms: V114, Schedule A: Participants 7-11 months; V114, Schedule B: Participants 12-23 months; V114, Schedule C: Participants 2-17 years
Biological: Prevnar 13® — Prevnar 13® 13-valent PCV containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) in each 0.5 mL IM administration.
  Other Names: PCV13
  Arms: Prevnar 13®, Schedule A: Participants 7-11 months; Prevnar 13®, Schedule B: Participants 12-23 months; Prevnar 13®, Schedule C: Participants 2-17 years

SUMMARY:
The purpose of this study is 1) to evaluate the safety and tolerability of V114 with respect to the proportion of participants with adverse events (AEs) and 2) to evaluate the anti-pneumococcal polysaccharide (PnPs) serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) at 30 days following the last dose for each vaccination group. There is no formal hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria

* Not be pregnant or breastfeeding
* Not be a woman of childbearing potential
* If of a woman of childbearing potential, agree to follow the contraceptive guidance during the treatment period and for at least 6 weeks after the last dose of study intervention
* Has a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent

Exclusion Criteria

* History of invasive pneumococcal disease (IPD)
* Known hypersensitivity to any component of the PCV or any diphtheria toxoid-containing vaccine
* Had a recent febrile illness occurring within 72 hours prior to receipt of study vaccine
* Known or suspected impairment of immunological function
* History of congenital or acquired immunodeficiency
* Has or his/her mother has a documented human immunodeficiency virus (HIV) infection
* Known or history of functional or anatomic asplenia
* Has failure to thrive based on the clinical judgement of the investigator
* Has a bleeding disorder contraindicating intramuscular vaccination
* Has a history of autoimmune disease (including but not limited to systemic lupus erythematosus, antiphospholipid syndrome, Behcet's disease, autoimmune thyroid disease, polymyositis and dermatomyositis, scleroderma, type 1 diabetes mellitus, or other autoimmune disorders)
* Has known neurologic or cognitive behavioral disorder, including encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive development disorder, and related disorders
* Is 7 to 23 months of age and has received a dose of a pneumococcal vaccine prior to study entry based on medical record. Participants ≥2 years of age could have received a PCV at least 8 weeks prior to study entry as follows: a partial regimen of Prevnar™,Synflorix™, or Prevnar 13™ or a full regimen of Prevnar™ or Synflorix™ based on local guidelines. Participants should not have received any dose of a pneumococcal polysaccharide vaccine
* Meets one or more of the following systemic corticosteroid exclusion criteria: has received systemic corticosteroids (equivalent of ≥2 mg/kg total daily dose of prednisone or ≥20 mg/day for persons weighing >10 kg) for ≥14 consecutive days and has not completed this course of treatment at least 30 days prior to the first dose of study vaccine at randomization; has received or is expected to receive systemic corticosteroids exceeding physiologic replacement doses (approximately 5 mg/day prednisone equivalent) within 14 days prior to any dose of study vaccine; or is expected to require systemic corticosteroids within 30 days after any study vaccination during conduct of the study (Note: Topical, ophthalmic and inhaled steroids are permitted)
* Has received other licensed non-live vaccines within 14 days before receipt of study vaccine. Exception: Inactivated influenza vaccine may be administered but must be given at least 7 days before receipt of study vaccine or at least 15 days after receipt of study vaccine
* Has received a licensed live vaccine within 30 days before receipt of study vaccine
* Has received a blood transfusion or blood products, including immunoglobulins, within 6 months before receipt of study vaccine
* Has participated in another clinical study of an investigational product before the beginning or anytime during the duration of the current clinical study

Ages: 7 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 606 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Merck Sharp & Dohme LLC
Locations (26):
- Finland (10):
  - Tampereen yliopisto Espoon rokotetutkimusklinikka ( Site 0007), Espoo
  - Tampereen yliopisto Etelä-Helsingin rokotetutkimusklinikka ( Site 0005), Helsinki
  - Tampereen yliopisto Ita-Helsingin rokotetutkimusklinikka ( Site 0006), Helsinki
  - Tampereen yliopisto Järvenpään rokotetutkimusklinikka ( Site 0003), Jarvenpaa
  - Tampereen yliopisto Kokkolan rokotetutkimusklinikka ( Site 0009), Kokkola
  - Tampereen yliopisto Oulun rokotetutkimusklinikka ( Site 0004), Oulu
  - Tampereen yliopisto Porin rokotetutkimusklinikka ( Site 0008), Pori
  - Seinajoki Vaccine Research Center ( Site 0010), Seinäjoki
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 0001), Tampere
  - Tampereen yliopisto Turun rokotetutkimusklinikka ( Site 0002), Turku
- Malaysia (2):
  - Sabah Womens & Childrens Hospital ( Site 0902), Kota Kinabalu
  - University Malaya Medical Centre ( Site 0901), Kuala Lumpur
- Poland (6):
  - Przychodnia Vitamed Gaaj i Cichomski Spolka Jawna ( Site 0212), Bydgoszcz
  - Centrum Medyczne Pratia Bydgoszcz ( Site 0210), Bydgoszcz
  - Spec Zesp Opieki Zdrowotnej nad Matka i Dzieckiem w Poznaniu ( Site 0213), Poznan
  - NZ Lecznictwa Ambulatoryjnego - Michalkowice - Jarosz i Partnerzy ( Site 0211), Siemianowice Śląskie
  - Uniwersytecki Szpital Kliniczny ( Site 0207), Wroclaw
  - SPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 0209), Łomianki
- Russia (4):
  - Central Clinical Hospital of Russian Academy Science ( Site 0317), Moscow
  - Children s City Polyclinic No. 45 of the Nevsky District ( Site 0312), Saint Petersburg
  - Research Institute of Children Infections ( Site 0301), Saint Petersburg
  - MAI Childrens City Clinical Hospital 11 ( Site 0305), Yekaterinburg
- Thailand (4):
  - Chulalongkorn University ( Site 0601), Bangkok
  - Vaccine Trial Center Faculty of Tropical Medicine ( Site 0603), Bangkok
  - Siriraj Hospital ( Site 0600), Bangkok
  - Srinagarind Hospital ( Site 0602), Khonkaen

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Banniettis N, Wysocki J, Szenborn L, Phongsamart W, Pitisuttithum P, Ramet M, Richmond P, Shi Y, Dagan R, Good L, Papa M, Lupinacci R, McFetridge R, Tamms G, Churchill C, Musey L, Bickham K; V114-024 PNEU-PLAN study group. A phase III, multicenter, randomized, double-blind, active comparator-controlled study to evaluate the safety, tolerability, and immunogenicity of catch-up vaccination regimens of V114, a 15-valent pneumococcal conjugate vaccine, in healthy infants, children, and adolescents (PNEU-PLAN). Vaccine. 2022 Oct 19;40(44):6315-6325. doi: 10.1016/j.vaccine.2022.09.003. Epub 2022 Sep 21. PMID 36150974

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of approximately 600 participants were planned for enrollment. Randomization was stratified by age and pneumococcal conjugate vaccine (PCV) history.
Period: Overall Study
Arm/Group | V114, Schedule A: Participants 7-11 Months | Prevnar 13®, Schedule A: Participants 7-11 Months | V114, Schedule B: Participants 12-23 Months | Prevnar 13®, Schedule B: Participants 12-23 Months | V114, Schedule C: Participants 2-17 Years | Prevnar 13®, Schedule C: Participants 2-17 Years
Started | 64 | 64 | 62 | 64 | 177 | 175
PCV Dose 1 | 64 | 64 | 62 | 64 | 177 | 175
PCV Dose 2 | 63 | 64 | 62 | 64 | 0 | 0
PCV Dose 3 | 63 | 64 | 0 | 0 | 0 | 0
Completed | 63 | 64 | 62 | 64 | 177 | 175
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn by Parent/Guardian | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114, Schedule A: Participants 7-11 Months | Prevnar 13®, Schedule A: Participants 7-11 Months | V114, Schedule B: Participants 12-23 Months | Prevnar 13®, Schedule B: Participants 12-23 Months | V114, Schedule C: Participants 2-17 Years | Prevnar 13®, Schedule C: Participants 2-17 Years | Total
Number analyzed (Participants) | 64 | 64 | 62 | 64 | 177 | 175 | 606
Age, Customized [Count of Participants; unit: Participants]
  7-11 Months | 64 | 64 | 0 | 0 | 0 | 0 | 128
  12-23 Months | 0 | 0 | 62 | 64 | 0 | 0 | 126
  ≥2 to <6 Years | 0 | 0 | 0 | 0 | 114 | 112 | 226
  ≥6 to 17 Years | 0 | 0 | 0 | 0 | 63 | 63 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 30 | 38 | 85 | 83 | 298
  Male | 35 | 31 | 32 | 26 | 92 | 92 | 308
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 64 | 64 | 62 | 63 | 176 | 174 | 603
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 53 | 53 | 52 | 53 | 60 | 56 | 327
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 11 | 11 | 10 | 11 | 117 | 118 | 278
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration of Serotype-specific Immunoglobulin G - Schedule A: 7-11 Months
Description: The geometric mean concentration (GMC) of immunoglobulin G (IgG) serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13®; and two serotypes (22F and 33F) which are unique to V114 was determined. Sera from participants was used to measure vaccine-induced anti-pneumococcal polysaccharides (PnPs) serotype-specific IgG for all the 15 serotypes using pneumococcal electrochemiluminescence (PnECL) assay. The within-group 95% confidence intervals (CIs) were derived by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: 30 days post last vaccination
Population: The analysis population included all randomized participants without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114, Schedule A: Participants 7-11 Months | Prevnar 13®, Schedule A: Participants 7-11 Months
Number analyzed (Participants) | 64 | 64
μg/mL
  Serotype 1: number analyzed (Participants) | 60 | 59
  Serotype 1 | 2.47 [2.09 to 2.92] | 3.66 [2.98 to 4.50]
  Serotype 3: number analyzed (Participants) | 60 | 59
  Serotype 3 | 2.65 [2.30 to 3.05] | 1.71 [1.40 to 2.08]
  Serotype 4: number analyzed (Participants) | 60 | 59
  Serotype 4 | 2.21 [1.82 to 2.68] | 3.85 [3.12 to 4.76]
  Serotype 5: number analyzed (Participants) | 60 | 59
  Serotype 5 | 3.82 [3.14 to 4.63] | 4.56 [3.58 to 5.80]
  Serotype 6A: number analyzed (Participants) | 60 | 59
  Serotype 6A | 2.23 [1.71 to 2.91] | 4.30 [3.28 to 5.65]
  Serotype 6B: number analyzed (Participants) | 60 | 59
  Serotype 6B | 3.03 [2.41 to 3.82] | 4.17 [3.25 to 5.36]
  Serotype 7F: number analyzed (Participants) | 60 | 59
  Serotype 7F | 5.16 [4.27 to 6.23] | 6.42 [5.25 to 7.85]
  Serotype 9V: number analyzed (Participants) | 60 | 59
  Serotype 9V | 2.61 [2.09 to 3.26] | 3.59 [2.86 to 4.51]
  Serotype 14: number analyzed (Participants) | 60 | 59
  Serotype 14 | 9.62 [7.94 to 11.67] | 13.07 [10.40 to 16.42]
  Serotype 18C: number analyzed (Participants) | 60 | 59
  Serotype 18C | 3.45 [2.80 to 4.24] | 3.50 [2.75 to 4.45]
  Serotype 19A: number analyzed (Participants) | 60 | 59
  Serotype 19A | 4.59 [3.95 to 5.33] | 5.81 [4.92 to 6.85]
  Serotype 19F: number analyzed (Participants) | 60 | 59
  Serotype 19F | 3.49 [2.94 to 4.15] | 4.83 [4.03 to 5.79]
  Serotype 23F: number analyzed (Participants) | 60 | 59
  Serotype 23F | 2.62 [2.02 to 3.39] | 2.79 [2.10 to 3.69]
  Serotype 22F: number analyzed (Participants) | 60 | 58
  Serotype 22F | 9.04 [7.48 to 10.93] | 0.14 [0.10 to 0.19]
  Serotype 33F: number analyzed (Participants) | 60 | 59
  Serotype 33F | 3.37 [2.78 to 4.10] | 0.13 [0.10 to 0.16]

2. Primary Outcome: GMC of Serotype-specific IgG - Schedule B: 12-23 Months
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13®; and two serotypes (22F and 33F) which are unique to V114 was determined. Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for all the 15 serotypes using pneumococcal electrochemiluminescence (PnECL) assay. The within-group 95% CIs were derived by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: 30 days post last vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114, Schedule B: Participants 12-23 Months | Prevnar 13®, Schedule B: Participants 12-23 Months
Number analyzed (Participants) | 62 | 64
μg/mL
  Serotype 1: number analyzed (Participants) | 56 | 60
  Serotype 1 | 3.83 [3.07 to 4.77] | 4.20 [3.30 to 5.34]
  Serotype 3: number analyzed (Participants) | 56 | 60
  Serotype 3 | 2.96 [2.44 to 3.58] | 1.68 [1.29 to 2.20]
  Serotype 4: number analyzed (Participants) | 56 | 60
  Serotype 4 | 3.46 [2.67 to 4.50] | 4.89 [3.76 to 6.36]
  Serotype 5: number analyzed (Participants) | 56 | 60
  Serotype 5 | 3.39 [2.65 to 4.34] | 3.12 [2.52 to 3.88]
  Serotype 6A: number analyzed (Participants) | 56 | 60
  Serotype 6A | 2.05 [1.30 to 3.23] | 3.73 [2.64 to 5.29]
  Serotype 6B: number analyzed (Participants) | 56 | 60
  Serotype 6B | 2.69 [1.70 to 4.25] | 2.87 [1.92 to 4.30]
  Serotype 7F: number analyzed (Participants) | 56 | 60
  Serotype 7F | 4.80 [3.63 to 6.34] | 5.42 [4.30 to 6.82]
  Serotype 9V: number analyzed (Participants) | 56 | 60
  Serotype 9V | 2.48 [1.97 to 3.11] | 2.89 [2.21 to 3.78]
  Serotype 14: number analyzed (Participants) | 56 | 60
  Serotype 14 | 8.23 [6.19 to 10.94] | 8.30 [6.56 to 10.51]
  Serotype 18C: number analyzed (Participants) | 56 | 60
  Serotype 18C | 5.09 [3.98 to 6.52] | 3.68 [2.85 to 4.75]
  Serotype 19A: number analyzed (Participants) | 56 | 60
  Serotype 19A | 6.74 [5.29 to 8.60] | 5.87 [4.85 to 7.11]
  Serotype 19F: number analyzed (Participants) | 56 | 60
  Serotype 19F | 5.90 [4.69 to 7.43] | 5.92 [4.93 to 7.11]
  Serotype 23F: number analyzed (Participants) | 56 | 60
  Serotype 23F | 2.85 [1.99 to 4.07] | 2.18 [1.54 to 3.07]
  Serotype 22F: number analyzed (Participants) | 56 | 60
  Serotype 22F | 15.90 [12.16 to 20.78] | 0.12 [0.09 to 0.16]
  Serotype 33F: number analyzed (Participants) | 56 | 60
  Serotype 33F | 5.17 [3.96 to 6.74] | 0.15 [0.12 to 0.19]

3. Primary Outcome: GMC of Serotype-specific IgG - Schedule C: 2-17 Years
Description: as for outcome 2
Time Frame: 30 days post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114, Schedule C: Participants 2-17 Years | Prevnar 13®, Schedule C: Participants 2-17 Years
Number analyzed (Participants) | 177 | 175
μg/mL
  Serotype 1: number analyzed (Participants) | 162 | 162
  Serotype 1 | 3.00 [2.60 to 3.46] | 3.99 [3.48 to 4.58]
  Serotype 3: number analyzed (Participants) | 162 | 162
  Serotype 3 | 1.37 [1.19 to 1.58] | 1.03 [0.88 to 1.21]
  Serotype 4: number analyzed (Participants) | 162 | 162
  Serotype 4 | 2.53 [2.17 to 2.96] | 5.22 [4.52 to 6.03]
  Serotype 5: number analyzed (Participants) | 162 | 162
  Serotype 5 | 3.43 [2.89 to 4.07] | 4.24 [3.46 to 5.20]
  Serotype 6A: number analyzed (Participants) | 162 | 162
  Serotype 6A | 9.03 [7.07 to 11.53] | 8.81 [6.96 to 11.14]
  Serotype 6B: number analyzed (Participants) | 162 | 161
  Serotype 6B | 13.55 [10.52 to 17.46] | 10.51 [8.01 to 13.78]
  Serotype 7F: number analyzed (Participants) | 162 | 162
  Serotype 7F | 4.03 [3.46 to 4.70] | 4.63 [3.92 to 5.46]
  Serotype 9V: number analyzed (Participants) | 162 | 162
  Serotype 9V | 3.60 [3.06 to 4.24] | 4.35 [3.65 to 5.20]
  Serotype 14: number analyzed (Participants) | 162 | 162
  Serotype 14 | 9.21 [7.11 to 11.92] | 8.04 [6.24 to 10.36]
  Serotype 18C: number analyzed (Participants) | 162 | 162
  Serotype 18C | 7.16 [6.03 to 8.52] | 4.46 [3.76 to 5.30]
  Serotype 19A: number analyzed (Participants) | 162 | 162
  Serotype 19A | 10.99 [9.12 to 13.26] | 14.90 [12.23 to 18.16]
  Serotype 19F: number analyzed (Participants) | 162 | 162
  Serotype 19F | 8.95 [7.45 to 10.76] | 12.28 [10.07 to 14.97]
  Serotype 23F: number analyzed (Participants) | 162 | 162
  Serotype 23F | 5.36 [4.41 to 6.50] | 5.12 [4.12 to 6.37]
  Serotype 22F: number analyzed (Participants) | 162 | 159
  Serotype 22F | 14.99 [12.73 to 17.66] | 0.31 [0.24 to 0.38]
  Serotype 33F: number analyzed (Participants) | 162 | 160
  Serotype 33F | 4.89 [4.12 to 5.80] | 0.27 [0.22 to 0.32]

4. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events - Schedule A: 7-11 Months
Description: An adverse event (AE) is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. The parent/guardian of the participant recorded the presence of any vaccination report card (VRC)-prompted injection-site AEs that occurred in the 14 days after any vaccination. The percentage of participants with an injection-site AE prompted on the VRC (redness/erythema, hardness/induration, swelling, and pain) was summarized.
Time Frame: Up to 14 days post any vaccination
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule A: Participants 7-11 Months | Prevnar 13®, Schedule A: Participants 7-11 Months
Number analyzed (Participants) | 64 | 64
Percentage of Participants
  Redness/Erythema | 28.1 [17.6 to 40.8] | 34.4 [22.9 to 47.3]
  Hardness/Induration | 17.2 [8.9 to 28.7] | 14.1 [6.6 to 25.0]
  Pain | 18.8 [10.1 to 30.5] | 7.8 [2.6 to 17.3]
  Swelling | 18.8 [10.1 to 30.5] | 15.6 [7.8 to 26.9]

5. Primary Outcome: Percentage of Participants With Solicited Injection-site AEs - Schedule B: 12-23 Months
Description: An AE is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. The parent/guardian of the participant recorded the presence of any vaccination report card (VRC)-prompted injection-site AEs that occurred in the 14 days after any vaccination. The percentage of participants with an injection-site AE prompted on the VRC (redness/erythema, hardness/induration, swelling, and pain) was summarized.
Time Frame: Up to 14 days post any vaccination
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule B: Participants 12-23 Months | Prevnar 13®, Schedule B: Participants 12-23 Months
Number analyzed (Participants) | 62 | 64
Percentage of Participants
  Redness/Erythema | 21.0 [11.7 to 33.2] | 21.9 [12.5 to 34.0]
  Hardness/Induration | 8.1 [2.7 to 17.8] | 9.4 [3.5 to 19.3]
  Pain | 33.9 [22.3 to 47.0] | 23.4 [13.8 to 35.7]
  Swelling | 14.5 [6.9 to 25.8] | 12.5 [5.6 to 23.2]

6. Primary Outcome: Percentage of Participants With Solicited Injection-site AEs - Schedule C: 2-17 Years
Description: as for outcome 5
Time Frame: Up to 14 days post vaccination
Population: The analysis population included all randomized participants who received 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule C: Participants 2-17 Years | Prevnar 13®, Schedule C: Participants 2-17 Years
Number analyzed (Participants) | 177 | 175
Percentage of Participants
  Redness/Erythema | 19.2 [13.7 to 25.8] | 21.1 [15.3 to 27.9]
  Hardness/Induration | 6.8 [3.6 to 11.5] | 14.9 [9.9 to 21.0]
  Pain | 54.8 [47.2 to 62.3] | 56.6 [48.9 to 64.0]
  Swelling | 20.9 [15.2 to 27.6] | 24.0 [17.9 to 31.0]

7. Primary Outcome: Percentage of Participants With Solicited Systemic AEs - Schedule A: 7-11 Months
Description: An AE is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. The parent/guardian of the participant recorded the presence of any VRC-prompted systemic AEs that occurred in the 14 days after any vaccination. For participants 7 months to <3 years of age at enrollment, solicited systemic AEs include irritability, drowsiness/somnolence, appetite lost/decreased appetite, and hives or welts/urticaria. The percentage of participants with a systemic AE was summarized.
Time Frame: Up to 14 days post any vaccination
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule A: Participants 7-11 Months | Prevnar 13®, Schedule A: Participants 7-11 Months
Number analyzed (Participants) | 64 | 64
Percentage of Participants
  Appetite lost/Decreased appetite | 15.6 [7.8 to 26.9] | 18.8 [10.1 to 30.5]
  Irritability | 32.8 [21.6 to 45.7] | 43.8 [31.4 to 56.7]
  Drowsiness/Somnolence | 21.9 [12.5 to 34.0] | 15.6 [7.8 to 26.9]
  Hives or Welts/Urticaria | 1.6 [0.0 to 8.4] | 4.7 [1.0 to 13.1]

8. Primary Outcome: Percentage of Participants With Solicited Systemic AEs - Schedule B: 12-23 Months
Description: as for outcome 7
Time Frame: Up to 14 days post any vaccination
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule B: Participants 12-23 Months | Prevnar 13®, Schedule B: Participants 12-23 Months
Number analyzed (Participants) | 62 | 64
Percentage of Participants
  Appetite lost/Decreased appetite | 22.6 [12.9 to 35.0] | 18.8 [10.1 to 30.5]
  Irritability | 35.5 [23.7 to 48.7] | 21.9 [12.5 to 34.0]
  Drowsiness/Somnolence | 24.2 [14.2 to 36.7] | 17.2 [8.9 to 28.7]
  Hives or Welts/Urticaria | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

9. Primary Outcome: Percentage of Participants With Solicited Systemic AEs - Schedule C: 2-17 Years
Description: An AE is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. The parent/guardian of the participant recorded the presence of any VRC-prompted systemic AEs that occurred in the 14 days after any vaccination. For participants 7 months to <3 years of age at enrollment, solicited systemic AEs include irritability, drowsiness/somnolence, appetite lost/decreased appetite, and hives or welts/urticaria. For participants ≥3 years of age at enrollment, solicited systemic AEs include muscle pain/ myalgia, joint pain/arthralgia, headache, tiredness/fatigue, and hives or welts/urticaria. The percentage of participants with a systemic AE was summarized.
Time Frame: Up to 14 days post vaccination
Population: The analysis population included all randomized participants who received 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule C: Participants 2-17 Years | Prevnar 13®, Schedule C: Participants 2-17 Years
Number analyzed (Participants) | 177 | 175
Percentage of Participants
  Joint pain/arthralgia | 0.0 [0.0 to 2.1] | 1.7 [0.4 to 4.9]
  Appetite lost/Decreased appetite | 2.3 [0.6 to 5.7] | 2.9 [0.9 to 6.5]
  Tiredness/Fatigue | 15.8 [10.8 to 22.0] | 17.1 [11.9 to 23.6]
  Headache | 11.9 [7.5 to 17.6] | 13.7 [9.0 to 19.7]
  Irritability | 2.8 [0.9 to 6.5] | 4.0 [1.6 to 8.1]
  Muscle pain/Myalgia | 23.7 [17.7 to 30.7] | 16.6 [11.4 to 22.9]
  Drowsiness/Somnolence | 2.8 [0.9 to 6.5] | 2.9 [0.9 to 6.5]
  Hives or Welts/Urticaria | 1.1 [0.1 to 4.0] | 1.1 [0.1 to 4.1]

10. Primary Outcome: Percentage of Participants With at Least 1 Vaccine-related Serious Adverse Event - Schedule A: 7-11 Months
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. SAEs that are reported to be at least possibly related by the investigator to study vaccination will be summarized. Estimated within-group CIs are calculated based on the exact binomial method proposed by Clopper and Pearson and are provided in accordance with the statistical analysis plan.
Time Frame: Up to ~6 months post final vaccination
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule A: Participants 7-11 Months | Prevnar 13®, Schedule A: Participants 7-11 Months
Number analyzed (Participants) | 64 | 64
Percentage of Participants | 0.0 (0.0) [0.0 to 5.6] | 0.0 (0.0) [0.0 to 5.6]

11. Primary Outcome: Percentage of Participants With at Least 1 Vaccine-related SAE - Schedule B: 12-23 Months
Description: as for outcome 10
Time Frame: Up to ~6 months post final vaccination
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule B: Participants 12-23 Months | Prevnar 13®, Schedule B: Participants 12-23 Months
Number analyzed (Participants) | 62 | 64
Percentage of Participants | 0.0 (0.0) [0.0 to 5.8] | 0.0 (0.0) [0.0 to 5.6]

12. Primary Outcome: Percentage of Participants With at Least 1 Vaccine-related SAE - Schedule C: 2-17 Years
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. SAEs that are reported to be at least possibly related by the investigator to study vaccination will be summarized.
Time Frame: Up to ~6 months post vaccination
Population: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule C: Participants 2-17 Years | Prevnar 13®, Schedule C: Participants 2-17 Years
Number analyzed (Participants) | 177 | 175
Percentage of Participants | 0.0 (0.0) [0.0 to 2.1] | 0.0 (0.0) [0.0 to 2.1]

13. Secondary Outcome: Percentage of Participants Meeting Serotype-specific IgG Threshold Value of ≥0.35 μg/mL for Each of the 15 Serotypes - Schedule A: 7-11 Months
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for all the 15 serotypes using PnECL assay. The percentage that achieved the IgG threshold value of ≥0.35 μg/mL was summarized. Estimated within-group CIs are calculated based on the exact binomial method proposed by Clopper and Pearson and are provided in accordance with the statistical analysis plan.
Time Frame: 30 days post final vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule A: Participants 7-11 Months | Prevnar 13®, Schedule A: Participants 7-11 Months
Number analyzed (Participants) | 64 | 64
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 60 | 59
  Serotype 1 | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 3: number analyzed (Participants) | 60 | 59
  Serotype 3 | 100.0 [94.0 to 100.0] | 96.6 [88.3 to 99.6]
  Serotype 4: number analyzed (Participants) | 60 | 59
  Serotype 4 | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 5: number analyzed (Participants) | 60 | 59
  Serotype 5 | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 6A: number analyzed (Participants) | 60 | 59
  Serotype 6A | 95.0 [86.1 to 99.0] | 98.3 [90.9 to 100.0]
  Serotype 6B: number analyzed (Participants) | 60 | 59
  Serotype 6B | 96.7 [88.5 to 99.6] | 100.0 [93.9 to 100.0]
  Serotype 7F: number analyzed (Participants) | 60 | 59
  Serotype 7F | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 9V: number analyzed (Participants) | 60 | 59
  Serotype 9V | 98.3 [91.1 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 14: number analyzed (Participants) | 60 | 59
  Serotype 14 | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 18C: number analyzed (Participants) | 60 | 59
  Serotype 18C | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 19A: number analyzed (Participants) | 60 | 59
  Serotype 19A | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 19F: number analyzed (Participants) | 60 | 59
  Serotype 19F | 100.0 [94.0 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 23F: number analyzed (Participants) | 60 | 59
  Serotype 23F | 98.3 [91.1 to 100.0] | 100.0 [93.9 to 100.0]
  Serotype 22F: number analyzed (Participants) | 60 | 58
  Serotype 22F | 100.0 [94.0 to 100.0] | 13.8 [6.1 to 25.4]
  Serotype 33F: number analyzed (Participants) | 60 | 59
  Serotype 33F | 100.0 [94.0 to 100.0] | 11.9 [4.9 to 22.9]

14. Secondary Outcome: Percentage of Participants Meeting Serotype-specific IgG Threshold Value of ≥0.35 μg/mL for Each of the 15 Serotypes - Schedule B: 12-23 Months
Description: Sera from participants was used to measure vaccine-induced anti-PnPs serotype-specific IgG for all the 15 serotypes using PnECL assay. The percentage that achieved the IgG threshold value of ≥0.35 μg/mL was summarized. Estimated within-group CIs are calculated based on the exact binomial method proposed by Clopper and Pearson and are provided in accordance with the statistical analysis plan. The analysis population included all randomized participants without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint.
Time Frame: 30 days post final vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule B: Participants 12-23 Months | Prevnar 13®, Schedule B: Participants 12-23 Months
Number analyzed (Participants) | 62 | 64
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 56 | 60
  Serotype 1 | 100.0 [93.6 to 100.0] | 98.3 [91.1 to 100.0]
  Serotype 3 (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 3 (n=56,60) | 98.2 [90.4 to 100.0] | 90.0 [79.5 to 96.2]
  Serotype 4 (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 4 (n=56,60) | 100.0 [93.6 to 100.0] | 96.7 [88.5 to 99.6]
  Serotype 5 (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 5 (n=56,60) | 98.2 [90.4 to 100.0] | 98.3 [91.1 to 100.0]
  Serotype 6A (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 6A (n=56,60) | 83.9 [71.7 to 92.4] | 95.0 [86.1 to 99.0]
  Serotype 6B (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 6B (n=56,60) | 89.3 [78.1 to 96.0] | 88.3 [77.4 to 95.2]
  Serotype 7F (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 7F (n=56,60) | 98.2 [90.4 to 100.0] | 100.0 [94.0 to 100.0]
  Serotype 9V (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 9V (n=56,60) | 98.2 [90.4 to 100.0] | 96.7 [88.5 to 99.6]
  Serotype 14 (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 14 (n=56,60) | 98.2 [90.4 to 100.0] | 100.0 [94.0 to 100.0]
  Serotype 18C (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 18C (n=56,60) | 96.4 [87.7 to 99.6] | 98.3 [91.1 to 100.0]
  Serotype 19A (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 19A (n=56,60) | 98.2 [90.4 to 100.0] | 100.0 [94.0 to 100.0]
  Serotype 19F (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 19F (n=56,60) | 100.0 [93.6 to 100.0] | 100.0 [94.0 to 100.0]
  Serotype 23F (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 23F (n=56,60) | 94.6 [85.1 to 98.9] | 88.3 [77.4 to 95.2]
  Serotype 22F (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 22F (n=56,60) | 100.0 [93.6 to 100.0] | 6.7 [1.8 to 16.2]
  Serotype 33F (n=56,60): number analyzed (Participants) | 56 | 60
  Serotype 33F (n=56,60) | 94.6 [85.1 to 98.9] | 15.0 [7.1 to 26.6]

15. Secondary Outcome: Percentage of Participants Meeting Serotype-specific IgG Threshold Value of ≥0.35 μg/mL for Each of the 15 Serotypes - Schedule C: 2-17 Years
Description: as for outcome 13
Time Frame: 30 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114, Schedule C: Participants 2-17 Years | Prevnar 13®, Schedule C: Participants 2-17 Years
Number analyzed (Participants) | 177 | 175
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 162 | 162
  Serotype 1 | 99.4 [96.6 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 3: number analyzed (Participants) | 162 | 162
  Serotype 3 | 95.7 [91.3 to 98.2] | 87.7 [81.6 to 92.3]
  Serotype 4: number analyzed (Participants) | 162 | 162
  Serotype 4 | 98.8 [95.6 to 99.9] | 100.0 [97.7 to 100.0]
  Serotype 5: number analyzed (Participants) | 162 | 162
  Serotype 5 | 99.4 [96.6 to 100.0] | 99.4 [96.6 to 100.0]
  Serotype 6A: number analyzed (Participants) | 162 | 162
  Serotype 6A | 98.1 [94.7 to 99.6] | 98.1 [94.7 to 99.6]
  Serotype 6B: number analyzed (Participants) | 162 | 162
  Serotype 6B | 98.1 [94.7 to 99.6] | 96.9 [92.9 to 99.0]
  Serotype 7F: number analyzed (Participants) | 162 | 162
  Serotype 7F | 99.4 [96.6 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 9V: number analyzed (Participants) | 162 | 162
  Serotype 9V | 100.0 [97.7 to 100.0] | 98.8 [95.6 to 99.9]
  Serotype 14: number analyzed (Participants) | 162 | 162
  Serotype 14 | 99.4 [96.6 to 100.0] | 98.1 [94.7 to 99.6]
  Serotype 18C: number analyzed (Participants) | 162 | 162
  Serotype 18C | 100.0 [97.7 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 19A: number analyzed (Participants) | 162 | 162
  Serotype 19A | 100.0 [97.7 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 19F: number analyzed (Participants) | 162 | 162
  Serotype 19F | 99.4 [96.6 to 100.0] | 100.0 [97.7 to 100.0]
  Serotype 23F: number analyzed (Participants) | 162 | 162
  Serotype 23F | 99.4 [96.6 to 100.0] | 95.7 [91.3 to 98.2]
  Serotype 22F: number analyzed (Participants) | 162 | 159
  Serotype 22F | 100.0 [97.7 to 100.0] | 37.7 [30.2 to 45.8]
  Serotype 33F: number analyzed (Participants) | 162 | 160
  Serotype 33F | 99.4 [96.6 to 100.0] | 37.5 [30.0 to 45.5]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: Up to 14 days after any vaccination; Serious adverse events and all-cause mortality: Up to ~6 months after the last vaccination.
Description: The analysis population included all randomized participants who received at least 1 dose of study intervention.
Groups:
- V114 (7-11 Months): Each participant received a 0.5 mL intramuscular (IM) injection for 7 to 11 months of age (Pneumococcal conjugate vaccine [PCV]-naïve). 3 doses. Dose 1: at randomization, Dose 2: 4 to 8 weeks after Dose 1, and Dose 3: 8 to 12 weeks after Dose 2 and ≥12 months of age.
- Prevnar (7-11 Months): Each participant received a 0.5 mL IM injection for 7 to 11 months of age (PCV-naïve). 3 doses. Dose 1: at randomization, Dose 2: 4 to 8 weeks after Dose 1, and Dose 3: 8 to 12 weeks after Dose 2 and ≥12 months of age.
- V114 (12-23 Months); Prevnar (12-23 Months): Each participant received a 0.5 mL IM injection for 12 to 23 months of age (PCV-naïve), 2 doses: Dose 1: at randomization, and Dose 2: 8 to 12 weeks after Dose 1.
- V114 (2-17 Years): Each participant received a 0.5 mL IM injection for 2 to 17 years of age (PCV-naïve or PCV experienced): Single dose administered at randomization and at least 8 weeks after previous PCV for participants who were PCV-experienced.
- Prevnar (2-17 Years): Each participant received a 0.5 mL IM injection for 2 to 17 years of age (PCV-naïve or PCV-experienced): Single dose administered at randomization and at least 8 weeks after previous PCV for participants who were PCV-experienced.
Arm/Group | V114 (7-11 Months) | Prevnar (7-11 Months) | V114 (12-23 Months) | Prevnar (12-23 Months) | V114 (2-17 Years) | Prevnar (2-17 Years)
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64 | 0/62 | 0/64 | 0/177 | 0/175
Serious Adverse Events (participants affected / at risk) | 7/64 | 5/64 | 4/62 | 4/64 | 4/177 | 4/175
Other Adverse Events (participants affected / at risk) | 44/64 | 47/64 | 46/62 | 36/64 | 125/177 | 125/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (7-11 Months) (N=64) | Prevnar (7-11 Months) (N=64) | V114 (12-23 Months) (N=62) | Prevnar (12-23 Months) (N=64) | V114 (2-17 Years) (N=177) | Prevnar (2-17 Years) (N=175)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (7-11 Months) (N=64) | Prevnar (7-11 Months) (N=64) | V114 (12-23 Months) (N=62) | Prevnar (12-23 Months) (N=64) | V114 (2-17 Years) (N=177) | Prevnar (2-17 Years) (N=175)
Injection site erythema (General disorders) | 18 (29) | 22 (36) | 13 (14) | 14 (16) | 34 (37) | 37 (37)
Injection site induration (General disorders) | 11 (20) | 9 (16) | 5 (8) | 6 (9) | 12 (13) | 26 (28)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 12 (23) | 10 (17) | 9 (11) | 8 (8) | 37 (39) | 42 (43)
Pyrexia (General disorders) | 20 (26) | 14 (16) | 9 (11) | 7 (7) | 13 (14) | 13 (14)
Injection site pain (General disorders) | 12 (19) | 5 (6) | 21 (27) | 15 (17) | 97 (111) | 99 (106)
Somnolence (Nervous system disorders) | 14 (22) | 10 (15) | 15 (29) | 11 (11) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 28 (42) | 30 (38)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 42 (46) | 30 (34)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 21 (32) | 24 (33)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (7) | 8 (11) | 7 (7) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 10 (15) | 12 (17) | 14 (21) | 12 (19) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 21 (39) | 28 (41) | 22 (33) | 14 (18) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT03885934/Prot_SAP_000.pdf